CLINICAL TRIAL: NCT01816932
Title: Home or Office Visit for Insertion of Etonogestrel Implant: A Pilot Study
Brief Title: Home or Office Visit for the Insertion of Implantable Birth Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Suji Uhm, MD/MPH Student, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01-13-41
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Contraception
MeSH Terms: interventions — House Calls; Office Visits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Visit (Experimental): 20 participants will be randomized to receive a home visit for the insertion of their implantable birth control rather than the standard office visit.
  Interventions: Procedure: Home Visit
- Office Visit (Placebo Comparator): 20 participants will be randomized to receive an office visit (standard of care).
  Interventions: Procedure: Office visit

INTERVENTIONS:
Procedure: Home Visit — The intervention is the location of the insertion visit.
  Arms: Home Visit
Procedure: Office visit
  Other Names: Placebo
  Arms: Office Visit

SUMMARY:
This is a pilot study in which women who desire an etonogestrel implant will be randomized to either a home or office insertion visit. The purpose of this research is to study the interest in, feasibility of, and rates of insertion for implantable birth control (Implanon®/Nexplanon®) when inserted at home visit appointments compared to standard office visit appointments.

The ultimate goal of the study is to reduce barriers to insertion of the etonogestrel implant and increase consistent and correct contraception use by introducing a previously unexplored method of access, the home visit.

ELIGIBILITY:
Inclusion criteria

* Women aged 18 and over
* Was pregnant within the last 10 weeks
* Interested in using the etonogestrel implant for contraception
* Willing to have investigators come to the home for an insertion visit
* Presenting to University Hospitals for delivery or contraception.
* Has running water and a working bathroom in the home
* Has a safe and private location in the home for the implant to be inserted

Exclusion criteria

* Current or history of thrombosis or thromboembolic disorders
* Liver tumors or active liver disease
* Undiagnosed abnormal genital bleeding
* Known or suspected breast cancer or history of breast cancer
* Allergic reaction to components (ethylene vinylacetate, etonogestrel, barium sulfate) of etonogestrel implant or local anesthetics
* Women currently taking hepatic enzyme inducers including but not exclusive to barbiturates, bosentan, carbamazepine, felbamate, griseofulvin, oxcarbazepine, phenylbutazone, phenytoin, rifampin, topiramate, protease inhibitors, and St. John's wort
* Uncontrolled hypertension
* Housing located greater than 10 miles from University Hospitals Center for Women's Health
* The location of the home is in a place that would not be safe for investigators
* Participant is homeless

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Insertion rates of implantable birth control | Two weeks post-implant insertion at the follow-up telephone call
  Assess rates of insertion of etonogestrel contraceptive implant in women randomly assigned to home visits or standard office visits.

SECONDARY OUTCOMES:
Interest in home visit option | Within 6-8 weeks of enrollment
  Questionnaires will be distributed at enrollment (Enrollment Questionnaire) and at the insertion visit (Post-Implant Insertion Questionnaire)
Rates of return for postpartum follow-up | Within 6-8 weeks of enrollment
  Data will be collected via electronic medical records to assess if women returned to clinic for their scheduled postpartum visits.

CONTACTS AND LOCATIONS:
Overall Officials: Suji Uhm, B.S., Principal Investigator — Case Western Reserve University; Lisa Perriera, M.D./M.P.H., Study Director — University Hospitals
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

REFERENCES:
- [Background] Finer LB, Henshaw SK. Disparities in rates of unintended pregnancy in the United States, 1994 and 2001. Perspect Sex Reprod Health. 2006 Jun;38(2):90-6. doi: 10.1363/psrh.38.090.06. PMID 16772190
- [Background] Singh S, Sedgh G, Hussain R. Unintended pregnancy: worldwide levels, trends, and outcomes. Stud Fam Plann. 2010 Dec;41(4):241-50. doi: 10.1111/j.1728-4465.2010.00250.x. PMID 21465725
- [Background] Gold RB, Sonfield A, Richards CL and Frost JJ. Next Steps for America's Family Planning Program: Leveraging the Potential of Medicaid and Title X in an Evolving Health Care System. <http://www.guttmacher.org/pubs/NextSteps.pdf>. New York: Guttmacher Institute, 2009.
- [Background] Kershaw TS, Niccolai LM, Ickovics JR, Lewis JB, Meade CS, Ethier KA. Short and long-term impact of adolescent pregnancy on postpartum contraceptive use: implications for prevention of repeat pregnancy. J Adolesc Health. 2003 Nov;33(5):359-68. doi: 10.1016/s1054-139x(03)00138-1. PMID 14596957
- [Background] Templeman CL, Cook V, Goldsmith LJ, Powell J, Hertweck SP. Postpartum contraceptive use among adolescent mothers. Obstet Gynecol. 2000 May;95(5):770-6. doi: 10.1016/s0029-7844(00)00787-0. PMID 10775745
- [Background] Shulman JJ, Merritt CG. Postpartum contraception: subsequent pregnancy, delivery, and abortion rates. Fertil Steril. 1976 Jan;27(1):97-103. PMID 1245250
- [Background] Ogburn JA, Espey E, Stonehocker J. Barriers to intrauterine device insertion in postpartum women. Contraception. 2005 Dec;72(6):426-9. doi: 10.1016/j.contraception.2005.05.016. Epub 2005 Aug 9. PMID 16307964
- [Background] Jackson RA, Schwarz EB, Freedman L, Darney P. Advance supply of emergency contraception. effect on use and usual contraception--a randomized trial. Obstet Gynecol. 2003 Jul;102(1):8-16. doi: 10.1016/s0029-7844(03)00478-2. PMID 12850599
- [Background] Chandra A, Martinez GM, Mosher WD, Abma JC, Jones J. Fertility, family planning, and reproductive health of U.S. women: data from the 2002 National Survey of Family Growth. Vital Health Stat 23. 2005 Dec;(25):1-160. PMID 16532609
- [Background] Zhu BP, Rolfs RT, Nangle BE, Horan JM. Effect of the interval between pregnancies on perinatal outcomes. N Engl J Med. 1999 Feb 25;340(8):589-94. doi: 10.1056/NEJM199902253400801. PMID 10029642
- [Background] Zilberman B. [Influence of short interpregnancy interval on pregnancy outcomes]. Harefuah. 2007 Jan;146(1):42-7, 78. Hebrew. PMID 17294848
- [Background] Frost JJ, Singh S, Finer LB. Factors associated with contraceptive use and nonuse, United States, 2004. Perspect Sex Reprod Health. 2007 Jun;39(2):90-9. doi: 10.1363/3909007. PMID 17565622
- [Background] Sable MR, Libbus MK, Chiu JE. Factors affecting contraceptive use in women seeking pregnancy tests: Missouri, 1997. Fam Plann Perspect. 2000 May-Jun;32(3):124-31. PMID 10894258
- [Background] Sable MR, Libbus MK. Beliefs concerning contraceptive acquisition and use among low-income women. J Health Care Poor Underserved. 1998 Aug;9(3):262-75. doi: 10.1353/hpu.2010.0467. PMID 10073208
- [Background] Radecki SE, Bernstein GS. Use of clinic versus private family planning care by low-income women: access, cost, and patient satisfaction. Am J Public Health. 1989 Jun;79(6):692-7. doi: 10.2105/ajph.79.6.692. PMID 2729465
- [Background] Silverman J, Torres A, Forrest JD. Barriers to contraceptive services. Fam Plann Perspect. 1987 May-Jun;19(3):94-7, 101-2. PMID 3622744
- [Background] Frost JJ, Darroch JE. Factors associated with contraceptive choice and inconsistent method use, United States, 2004. Perspect Sex Reprod Health. 2008 Jun;40(2):94-104. doi: 10.1363/4009408. PMID 18577142
- [Background] Hatcher RA, Trussell J, Nelson AL, Cates W Jr, Stewart F, Kowal D, editors. Contraceptive technology. 19th rev. ed. New York (NY): Ardent Media, Inc.; 2007.
- [Background] Mosher WD, Jones J. Use of contraception in the United States: 1982-2008. Vital Health Stat 23. 2010 Aug;(29):1-44. PMID 20939159
- [Background] Harper CC, Blum M, de Bocanegra HT, Darney PD, Speidel JJ, Policar M, Drey EA. Challenges in translating evidence to practice: the provision of intrauterine contraception. Obstet Gynecol. 2008 Jun;111(6):1359-69. doi: 10.1097/AOG.0b013e318173fd83. PMID 18515520
- [Background] Madden T, Allsworth JE, Hladky KJ, Secura GM, Peipert JF. Intrauterine contraception in Saint Louis: a survey of obstetrician and gynecologists' knowledge and attitudes. Contraception. 2010 Feb;81(2):112-6. doi: 10.1016/j.contraception.2009.08.002. Epub 2009 Sep 16. PMID 20103447
- [Background] Trussell J, Lalla AM, Doan QV, Reyes E, Pinto L, Gricar J. Cost effectiveness of contraceptives in the United States. Contraception. 2009 Jan;79(1):5-14. doi: 10.1016/j.contraception.2008.08.003. Epub 2008 Sep 25. PMID 19041435
- [Background] Secura GM, Allsworth JE, Madden T, Mullersman JL, Peipert JF. The Contraceptive CHOICE Project: reducing barriers to long-acting reversible contraception. Am J Obstet Gynecol. 2010 Aug;203(2):115.e1-7. doi: 10.1016/j.ajog.2010.04.017. Epub 2010 Jun 11. PMID 20541171
- [Background] ACOG Practice Bulletin No. 121: Long-acting reversible contraception: Implants and intrauterine devices. Obstet Gynecol. 2011 Jul;118(1):184-196. doi: 10.1097/AOG.0b013e318227f05e. No abstract available. PMID 21691183
- [Background] Peipert JF, Zhao Q, Allsworth JE, Petrosky E, Madden T, Eisenberg D, Secura G. Continuation and satisfaction of reversible contraception. Obstet Gynecol. 2011 May;117(5):1105-1113. doi: 10.1097/AOG.0b013e31821188ad. PMID 21508749
- [Background] Tocce KM, Sheeder JL, Teal SB. Rapid repeat pregnancy in adolescents: do immediate postpartum contraceptive implants make a difference? Am J Obstet Gynecol. 2012 Jun;206(6):481.e1-7. doi: 10.1016/j.ajog.2012.04.015. Epub 2012 Apr 16. PMID 22631865
- [Background] Tocce K, Sheeder J, Python J, Teal SB. Long acting reversible contraception in postpartum adolescents: early initiation of etonogestrel implant is superior to IUDs in the outpatient setting. J Pediatr Adolesc Gynecol. 2012 Feb;25(1):59-63. doi: 10.1016/j.jpag.2011.09.003. Epub 2011 Nov 3. PMID 22051792
- [Background] Melnick AL, Rdesinski RE, Creach ED, Choi D, Harvey SM. The influence of nurse home visits, including provision of 3 months of contraceptives and contraceptive counseling, on perceived barriers to contraceptive use and contraceptive use self-efficacy. Womens Health Issues. 2008 Nov-Dec;18(6):471-81. doi: 10.1016/j.whi.2008.07.011. Epub 2008 Oct 15. PMID 18926726
- [Background] Peipert JF, Madden T, Allsworth JE, Secura GM. Preventing unintended pregnancies by providing no-cost contraception. Obstet Gynecol. 2012 Dec;120(6):1291-7. doi: 10.1097/aog.0b013e318273eb56. PMID 23168752
- [Derived] Uhm S, Pope R, Schmidt A, Bazella C, Perriera L. Home or office etonogestrel implant insertion after pregnancy: a randomized trial. Contraception. 2016 Nov;94(5):567-571. doi: 10.1016/j.contraception.2016.06.018. Epub 2016 Jun 29. PMID 27373542